CLINICAL TRIAL: NCT03721627
Title: Efficacy and Safety of Ledipasvir/Sofosbuvir Fixed Dose Combination Therapy in Treatment of Chronic Hepatitis C Infection in Egyptian Children With Gaucher Disease
Brief Title: Chronic Hepatitis C Treatment in Egyptian Children With Gaucher Disease.
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mansoura University Children Hospital (Other)
Responsible Party: Principal Investigator, Ahmed Megahed, MD, Associate Professor of Pediatrics, Mansoura University Children Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: R.18.03.130.R1
Record Dates: First submitted 2018-10-25; First posted 2018-10-26 (Actual); Last update posted 2018-10-30 (Actual); Status verified 2018-10

CONDITIONS: Gaucher Disease; HCV
Keywords: Ledipasvir/Sofosbuvir; Gaucher disease; HCV
MeSH Terms: conditions — Gaucher Disease | interventions — ledipasvir, sofosbuvir drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment group (Experimental): Ledipasvir/sofosbuvir fixed dose combination tablet (90 mg ledipasvir, 400 mg sofosbuvir) once daily for 12 weeks for those 12-18 years, Wt 35 kg or more and half the dose (45 mg ledipasvir, 200 mg sofosbuvir) once daily for 12 weeks for those 6-11 years, Wt Less than 35 kg.
  Interventions: Drug: Ledipasvir/Sofosbuvir

INTERVENTIONS:
Drug: Ledipasvir/Sofosbuvir — Direct acting anti HCV drugs

SUMMARY:
This prospective open label study is designed to screen all available Gaucher disease patients [either on enzyme replacement therapy (ERT) or not] for hepatitis C virus (HCV) infection. Furthermore to evaluate the safety and effectiveness of combined Sofosbuvir/Ledipasvir regimen given for 12 weeks in chronically infected patients aged 6-18 years.

DETAILED DESCRIPTION:
This is a prospective open label study, all Gaucher disease pediatric patients (6-18 years), diagnosed at or referred to the HCV Egyptian treatment site, Mansoura University Children's Hospital Gastroenterology and hepatology unit, after positive HCV screen results by Anti HCV antibodies and confirmatory positive quantitative HCV polymerase chain reaction (PCR) are going to be enrolled. Study protocol had been approved by the Mansoura faculty of Medicine Institutional Review Board (IRB).

Study design: In this prospective study, patients will receive ledipasvir-sofosbuvir fixed dose combination tablet (90 mg ledipasvir, 400 mg sofosbuvir) once daily for 12 weeks for those 12-18 years and half the dose (45 mg ledipasvir, 200 mg sofosbuvir) once daily for 12 weeks for those 6-11 years. After the period of treatment, follow up visit are arranged at 4, 12 and 24 weeks post-treatment.

Methods:

Every patient will be subjected to the following:

A. History taking: time and route of acquisition, medications including previous antiviral therapy B. Comprehensive medical examination before study entry will be carried out for all participants and symptom-directed examination in every visit.

C. In every visit, adverse events and concurrent medication will be reported for safety issue.

D. Tanner staging for pubertal assessment will be done for all patients prior to enrollment then at the end of therapy and end of post-treatment follow up.

E. Laboratory tests: All patients had positive (Anti-HCV Ab) and HCV-RNA PCR for more than 6 months. HCV-RNA will be measured Basal pretreatment at week 12 on treatment then at week 12, 24 post-treatment. Complete blood count (CBC),liver function tests (LFTs), international normalized ratio (INR), and serum creatinine will be done in the same time frame. Lab investigations are going to be done as a part of the routine work, using commercially available kits.

F. Percutaneous liver biopsy: Histological examination of liver biopsy will be done for all patients when feasible (Hemoglobin more than 10gm/dl, Platlet count more than 100 x103/mm2, Prothrombin time (PT) less than 3 seconds prolongation) and agreed by the patients and legal guardians. Liver fibrosis and necroinflammatory injury are going to be reported by a single expert pathologist according to the Modified Knodell score by Ishak, in which inflammatory activity is graded from 0-18 and fibrosis is graded from 0-6. Alternatively transient hepatic elastography by fibroscan is going to be done for those patients with contraindication or refusing liver biopsy.

ELIGIBILITY:
Inclusion Criteria:

* Aged 6 to <18 years
* Parent or legal guardian must provide written informed consent
* Treatment naïve or experienced children with chronic HCV infection
* Chronic HCV infection (≥ 6 months) documented by medical history or liver biopsy
* Screening laboratory values within defined thresholds
* No History of solid organ or bone marrow transplantation
* No history of clinical hepatic decompensation (eg, ascites, jaundice, encephalopathy, variceal hemorrhage)

Exclusion Criteria:

* Patients with other sever comorbidities of chronic medical illness (e.g. decompensated heart disease, chronic kidney insufficiency)
* Concomitant hepatitis B virus (HBV) or Human immunodeficiency virus (HIV) infection
* Medications (systemic steroids, immunosuppressives)
* Patients or guardians who are unwilling to participate or sign informed consent

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 10 (Estimated)
Dates: Start 2018-04-03 (Actual); Primary Completion 2019-04 (Estimated); Study Completion 2019-10 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients with Sustained Virologic Response | 18 months
  Proportion of patients achieving negative HCV PCR 12 weeks after therapy

SECONDARY OUTCOMES:
Prevalence of HCV infection among Gaucher disease children | 12 months
  Number of HCV PCR positive Gaucher disease patients/Number of screened Gaucher Disease patients
Drug intolerability | 18 months
  Proportion of patients who permanently discontinue study drug due to an adverse event.

CONTACTS AND LOCATIONS:
Locations (1):
- Mansoura University Children Hospital, Ped Gastroenteroloy and Hepatology Unit, Al Mansurah, Dakahliya, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Balistreri WF, Murray KF, Rosenthal P, Bansal S, Lin CH, Kersey K, Massetto B, Zhu Y, Kanwar B, German P, Svarovskaia E, Brainard DM, Wen J, Gonzalez-Peralta RP, Jonas MM, Schwarz K. The safety and effectiveness of ledipasvir-sofosbuvir in adolescents 12-17 years old with hepatitis C virus genotype 1 infection. Hepatology. 2017 Aug;66(2):371-378. doi: 10.1002/hep.28995. Epub 2017 Jun 19. PMID 27997679
- [Background] KF Murray, W Balistreri, S Bansal, et al. Ledipasvir/sofosbuvir ± ribavirin for 12 or 24 weeks is safe and effective in children 6-11 years old with chronic hepatitis C infection. EASL International Liver Congress. Amsterdam, April 19-23, 2017. Abstract GS-010.
- [Background] Adar T, Ilan Y, Elstein D, Zimran A. Liver involvement in Gaucher disease - Review and clinical approach. Blood Cells Mol Dis. 2018 Feb;68:66-73. doi: 10.1016/j.bcmd.2016.10.001. Epub 2016 Oct 19. PMID 27842801